CLINICAL TRIAL: NCT04405830
Title: Outcome of Patients Treated With Renal Replacement Therapy
Brief Title: Outcome of Patients Treated With RRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, : Investigator of Department of Cardiac Surgery, Nanjing Medical University
Other Study IDs: RRT-Jsph
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Acute Kidney Injury; Cardiac Surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Renal replacement therapy — Renal replacement therapy (RRT) refers to modalities of treatment that are used to replace the waste filtering functions of a normal kidney.

SUMMARY:
Acute Kidney Injury (AKI) is a common serious complication after cardiac surgery. AKI not only prolongs the hospitalization time of patients undergoing cardiac surgery and increases the cost of treatment, but also is an independent risk factor for postoperative death. The aim of this study is to investigate the outcome of patients treated with renal replacement therapy (RRT), and to evaluate the short-term and long-term outcomes of patients with RRT.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients undergoing cardiovascular surgery admitted to intensive care units.
* Patients receiving RRT for renal support
* Patients over 18 years of age

Exclusion Criteria:

* Patients <18 years
* Refusal of consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving RRT for renal support
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days after Renal replacement therapy

SECONDARY OUTCOMES:
ICU Length of Stay (LOS) | from ICU admission to ICU discharge, within 30 days of admission

CONTACTS AND LOCATIONS:
Overall Officials: Yong-feng Shao, MD, Study Director — First Hospital Affiliated to Nanjing Medical University
Locations (1):
- The first affiliated hospital of nanjing medical university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided